CLINICAL TRIAL: NCT07129915
Title: Effect of Nudge-Based Shared Decision Making on Self-Management Among Patients With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Nudge-Based Shared Decision Making and Self-Management in Type 2 Diabetes: A Randomized Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunxuan Li (Other)
Responsible Party: Sponsor-Investigator, Yunxuan Li, Principal Investigator and Graduate Student Researcher, School of Medicine, Xiamen University, Xiamen University
Organization: Xiamen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: XAHLL2025049
Record Dates: First submitted 2025-08-01; First posted 2025-08-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Physician-Patient Relations; Self-management
Keywords: Linguistic Nudging; Shared Decision Making; Randomized Controlled Trial; Mobile Health Application; Chinese Population
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linguistic Nudging Group (Experimental): Receives communication training + preference app
  Interventions: Behavioral: Linguistic Nudging Training; Device: Medication Preference App; Other: Standard Diabetes Care
- Standard Care Group (Other): Receives routine diabetes management only
  Interventions: Other: Standard Diabetes Care

INTERVENTIONS:
Behavioral: Linguistic Nudging Training — Physicians receive 4-hour communication training to optimize shared decision-making using behavioral nudging techniques
  Arms: Linguistic Nudging Group
Device: Medication Preference App — Patients use WeChat-based mini-program to record daily medication preferences and concerns
  Arms: Linguistic Nudging Group
Other: Standard Diabetes Care — Routine follow-up visits, HbA1c monitoring, and basic health education per hospital protocol

SUMMARY:
This study aims to test whether a communication strategy called "linguistic nudging" can help doctors and patients with type 2 diabetes make better treatment decisions together, and whether this improves patients' ability to manage their condition.

What will happen in the study? - 250 adults with type 2 diabetes from Xiang'an Hospital (Xiamen) will be randomly assigned to one of two groups:

Intervention group:Doctors will receive special training in "linguistic nudging" techniques to encourage shared decision-making. Patients will use a mobile app to record medication preferences, and doctors will adjust advice based on these preferences.

Control group:Patients will receive standard diabetes care without these additional strategies.

- All participants will be followed for 6 months.

What is the study aiming to find out?

The main goal is to see if patients in the intervention group:

Better follow medication plans Improve blood sugar monitoring Have better blood sugar control Feel more satisfied with doctor-patient communication

Why is this important? Good self-management is key to controlling diabetes, but many patients struggle with it. Effective communication during shared decision-making may empower patients to manage their condition day-to-day with greater confidence.

Patient safety and rights:

Participation is completely voluntary All personal information will be kept strictly confidential Medical support will be provided if any health problems occur during the study Participants may withdraw at any time

This research has been approved by the Ethics Committee of Xiang'an Hospital (Approval date: October 2025).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type 2 diabetes
* Age ≥ 18 years
* Normal cognitive function (assessed by Mini-Cog score ≥ 3)
* Basic smartphone operation ability (can independently use WeChat)
* Willing to participate and sign informed consent

Exclusion Criteria:

* Severe acute complications (e.g., ketoacidosis, hyperosmolar coma)
* Documented cognitive impairment (dementia, Alzheimer's, etc.)
* Currently participating in other clinical trials
* Life expectancy < 6 months
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) Level | Baseline and Month 6
  Absolute change in HbA1c (%) from baseline to 6 months, measured by high-performance liquid chromatography (HPLC). Reflects average blood glucose control over 3 months.
Diabetes Self-Management Capacity Scale Score | Baseline, Month 3, Month 6
  Composite score (0-100) based on validated 20-item scale assessing medication adherence, dietary control, physical activity, and blood glucose monitoring. Higher scores indicate better self-management capacity.
Shared Decision Making Questionnaire (SDM-Q-9) Score | Baseline
  Patient-reported evaluation of shared decision quality using 9-item Likert scale (0-45). Assesses physician-patient collaboration in treatment choices. Higher scores indicate better shared decision-making.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiang'an Hospital Affiliated to Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No